CLINICAL TRIAL: NCT07366554
Title: Exploration of Epigenetic Factors of Colorectal Adenoma in Korean
Brief Title: Epigenetic Factors of Colorectal Adenoma in Korean
Status: Not yet recruiting | Type: Observational
Sponsor: Bundang CHA Hospital (Other)
Responsible Party: Principal Investigator, KIM OneJoong, Clinical Assistant Professor, Bundang CHA Hospital
Other Study IDs: CHAMC IRB 2025-05-034-004
Record Dates: First submitted 2025-11-14; First posted 2026-01-26 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Adenoma; Colorectal Cancer Precancerous Lesion
Keywords: Colorectal Adenoma; DNA Methylation; Epigenetics; Biomarker discovery; SFRP2; TFPI2; SEPT9; SDC2; qMSP; Korean population; Colorectal cancer prevention; Adenoma-carcinoma sequence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Tissue, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal Adenoma Group: Participants undergoing colonoscopic polypectomy for colorectal adenoma. Adenomatous tissue and adjacent normal mucosa will be collected for methylation and sequencing analysis.

SUMMARY:
This study aims to explore epigenetic factors associated with colorectal adenoma (CRA) in the Korean population. CRA is a key precancerous lesion in the adenoma-carcinoma sequence, and identifying methylated genetic markers may improve early detection and risk stratification for colorectal cancer (CRC).

A total of 32 patients undergoing colonoscopic polypectomy will be enrolled. Adenomatous and adjacent normal tissues will be collected for deoxyribonucleic acid (DNA) extraction and bisulfite conversion. Quantitative methylation-specific polymerase chain reaction (qMSP) and Sanger sequencing will be used to assess the methylation status of candidate genes (SFRP2, TFPI2, SEPT9, and SDC2). Stool samples will also be analyzed by whole-genome sequencing (WGS) to evaluate microbiome and genetic profiles.

The study seeks to determine whether methylation levels of these genes are significantly elevated in adenoma tissue compared with normal mucosa, thereby identifying potential biomarkers for colorectal neoplasia surveillance and personalized colonoscopy follow-up intervals.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common malignancies in Korea, ranking second in national cancer incidence statistics. Most CRCs arise through the adenoma-carcinoma sequence, in which epigenetic and genetic alterations play critical roles. Identifying methylated genetic markers in colorectal adenoma may provide insights into early carcinogenic mechanisms and enable more individualized surveillance strategies after polypectomy.

This study focuses on exploring epigenetic factors-particularly DNA methylation patterns-associated with colorectal adenoma in Korean patients. A total of 32 participants undergoing colonoscopic polypectomy will be recruited. From each participant, both adenomatous tissue and adjacent normal mucosa (approximately 5 millimeters (mm) in size) will be collected. Stool samples will also be obtained for microbiome and genomic analysis.

DNA extracted from tissue and stool samples will undergo bisulfite conversion using the EZ DNA Methylation-Gold Kit (Zymo Research). Quantitative methylation-specific polymerase chain reaction (qMSP) will be performed to evaluate promoter methylation levels of four candidate genes-SFRP2 (Secreted Frizzled Related Protein 2), TFPI2 (Tissue Factor Pathway Inhibitor 2), SEPT9 (Septin 9), and SDC2 (Syndecan 2)-that have previously shown potential as colorectal neoplasia biomarkers. Selected samples will also undergo Sanger sequencing for CpG-level methylation profiling. Stool DNA will be analyzed through whole-genome sequencing (WGS) on the Illumina NovaSeq 6000 platform to assess microbial composition and genetic context.

Methylation indices (MtI) and percentage of methylated reference (PMR) values will be calculated and compared between adenoma and adjacent normal tissues. Receiver operating characteristic (ROC) curve analysis will determine the sensitivity and specificity of each gene as a potential biomarker.

By identifying methylated genes that are significantly upregulated in adenomatous tissues, this study aims to propose candidate epigenetic markers for predicting the recurrence or malignant transformation of colorectal adenoma. The findings may contribute to refining post-polypectomy surveillance intervals and supporting precision prevention strategies in CRC.

ELIGIBILITY:
* Inclusion Criteria:

  * Adults aged 19-85 years
  * Undergoing colonoscopic polypectomy for colorectal adenoma
  * Able to understand the study purpose and provide written informed consent
  * Adequate tissue available for both adenoma and adjacent normal mucosa sampling
* Exclusion Criteria:

  * History of colorectal cancer, inflammatory bowel disease, or hereditary colorectal cancer syndrome (e.g., FAP, Lynch syndrome)
  * Previous colorectal surgery that may alter anatomy or pathology
  * Inadequate sample quality or failure of DNA extraction
  * Refusal or withdrawal of informed consent
  * Severe comorbidities that make participation unsuitable at investigator's discretion

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing colonoscopic polypectomy for colorectal adenoma at Bundang CHA Hospital. Participants will be enrolled consecutively among those who provide written informed consent for collection of adenomatous and adjacent normal tissues. The study population represents adults aged 19-85 years who are clinically eligible for colonoscopy and tissue sampling
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-05-09 (Estimated); Study Completion 2027-05-09 (Estimated)

PRIMARY OUTCOMES:
Methylation index of SFRP2 in colorectal tissue | Baseline (Single Time Point)]
  Quantitative assessment of DNA methylation levels in adenomatous versus adjacent normal colorectal tissues. Methylation levels will be determined using quantitative methylation-specific PCR (qMSP) and expressed as methylation index (MtI, %).
Methylation index of TFPI2 in colorectal tissue | Baseline (Single Time Point)]
  Quantitative assessment of DNA methylation levels in adenomatous versus adjacent normal colorectal tissues. Methylation levels will be determined using quantitative methylation-specific PCR (qMSP) and expressed as methylation index (MtI, %).
Methylation index of SEPT9 in colorectal tissue | Baseline (Single Time Point)]
  Quantitative assessment of DNA methylation levels in adenomatous versus adjacent normal colorectal tissues. Methylation levels will be determined using quantitative methylation-specific PCR (qMSP) and expressed as methylation index (MtI, %).
Methylation index of SDC2 in colorectal tissue | Baseline (Single Time Point)]
  Quantitative assessment of DNA methylation levels in adenomatous versus adjacent normal colorectal tissues. Methylation levels will be determined using quantitative methylation-specific PCR (qMSP) and expressed as methylation index (MtI, %).

SECONDARY OUTCOMES:
Sensitivity and specificity of methylated SFRP2 for detecting adenoma | Baseline (Single Time Point)
  Receiver operating characteristic (ROC) curve analysis will be used to evaluate the diagnostic performance of methylated SFRP2 in distinguishing adenomatous from normal tissue. The percentage of methylated reference (PMR) values derived from qMSP will be compared between groups.
Sensitivity and specificity of methylated TFPI2 for detecting adenoma | Baseline (Single Time Point)
  Receiver operating characteristic (ROC) curve analysis will be used to evaluate the diagnostic performance of methylated TFPI2 in distinguishing adenomatous from normal tissue. The percentage of methylated reference (PMR) values derived from qMSP will be compared between groups.
Sensitivity and specificity of methylated SEPT9 for detecting adenoma | Baseline (Single Time Point)
  Receiver operating characteristic (ROC) curve analysis will be used to evaluate the diagnostic performance of methylated SEPT9 in distinguishing adenomatous from normal tissue. The percentage of methylated reference (PMR) values derived from qMSP will be compared between groups.
Sensitivity and specificity of methylated SDC2 for detecting adenoma | Baseline (Single Time Point)
  Receiver operating characteristic (ROC) curve analysis will be used to evaluate the diagnostic performance of methylated SDC2 in distinguishing adenomatous from normal tissue. The percentage of methylated reference (PMR) values derived from qMSP will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Bundang CHA Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2025-07-02): https://cdn.clinicaltrials.gov/large-docs/54/NCT07366554/Prot_ICF_000.pdf